CLINICAL TRIAL: NCT06214481
Title: A Phase 1, Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Rocatinlimab (AMG 451) Administered Subcutaneously in Healthy Chinese Subjects
Brief Title: A Study to Evaluate Rocatinlimab (AMG 451) in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20210186
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; AMG 451; KHK4083; Rocatinlimab
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rocatinlimab (Experimental): Participants will receive a single SC dose of rocatinlimab.
  Interventions: Drug: Rocatinlimab

INTERVENTIONS:
Drug: Rocatinlimab — Administered SC.
  Other Names: AMG 451

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetics of rocatinlimab after single subcutaneous (SC) administration in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a resident in mainland China, and of Chinese ancestry (participants whose parents within 3 generations are of Chinese ancestry).
* Healthy male or female participants, between 18 and 65 years of age (inclusive) at the time of screening.
* Body mass index between 18 and 30 kg/m^2 (inclusive) at the time of screening and check-in.
* Provide signed informed consent.

Exclusion Criteria:

* History or evidence, at screening or check-in, of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* Evidence of any active bacterial, viral, or fungal infection at screening including but not limited to upper or lower respiratory tract infection, conjunctivitis, acute otitis media, gastritis, enteritis, skin infections, infections requiring treatment with systemic therapy (antibiotics, antiviral, antiparasitic, antiprotozoal, or antifungals) for which therapy has not been completed within 4 weeks before enrollment.
* Immunocompromised participants at risk for viral reactivation including participants with history of solid organ transplantation, hematopoietic stem cell transplantation, or cellular therapy.
* Participants with disrupted skin integrity (apparent burn or dermatitis).
* Prior history of autoimmune disease including but not limited to inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), lupus, rheumatoid arthritis, psoriasis/psoriatic arthritis, multiple sclerosis.
* Positive hepatitis B surface antigen (HBsAg)/hepatitis B core antibody (HBcAb) or hepatitis C virus antibody and/or positive human immunodeficiency virus test, at screening. Participants whose hepatitis B and C results are compatible with prior immunity (resulting from inoculation) may be included.
* Positive T-spot test at screening.
* Participants who have received live vaccines within 5 weeks prior to screening, or plan to receive live vaccines within 120 days after administration of an investigational product.
* Participants who have received coronavirus disease 2019 vaccine within 30 days prior to check-in, or plan to receive a coronavirus disease 2019 vaccine within 120 days post-dose.
* Use of any over-the-counter or prescription medications within 30 days or 5 half-lives (whichever is longer) before check-in.

  1. Acetaminophen (paracetamol; up to 2 g/day) for analgesia will be allowed.
  2. Hormone replacement therapy (e.g., estrogen) and hormonal contraceptives will be allowed.
* Participant has received a dose of an investigational drug within the past 90 days or 5 half-lives, whichever is longer, prior to check-in.
* Have previously completed or withdrawn from this study or any other study investigating rocatinlimab or have previously received the investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Rocatinlimab | Up to day 126
Area Under the Serum Concentration Time Curve (AUC) from Time Zero to the Time of the Last Measurable Concentration (AUClast) of Rocatinlimab | Up to day 126
AUC from Time Zero to Infinity (AUCinf) of Rocatinlimab | Up to day 126

SECONDARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events | Up to day 126
Number of Participants Experiencing Serious Adverse Events | Up to day 126
Number of Participants who Develop Anti-rocatinlimab Antibodies | Up to day 126

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Huashan Hospital Affiliated to Fudan University?, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com